CLINICAL TRIAL: NCT00493181
Title: The Effect of Interleukin 11 on Thrombocytopenia Associated With Imatinib or Other Tyrosine Kinase Inhibitor Therapy in Patients With Chronic Myelogenous Leukemia
Brief Title: Interleukin 11, Thrombocytopenia, Imatinib in Chronic Myelogenous Leukemia (CML) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0113
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Results first posted 2011-05-04 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Leukemia; Chronic Myelogenous Leukemia; Chronic Myeloid Leukemia
Keywords: oprelvekin; tyrosine kinase inhibitor; Chronic Myelogenous Leukemia; Leukemia; CML; Thrombocytopenia; Imatinib; IL-11; Interleukin 11; Neumega
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Thrombocytopenia | interventions — Interleukin-11; oprelvekin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interleukin-11 (Experimental): Starting dose 10 mcg/kg subcutaneously 3 times a week
  Interventions: Drug: Interleukin-11 (IL-11 or Neumega)

INTERVENTIONS:
Drug: Interleukin-11 (IL-11 or Neumega) — 10 mcg/kg under the skin (usually of the arms, legs or abdomen) three times weekly. If the treatment is well tolerated but there is not enough of a platelet improvement, the dose and frequency of injections may be increased.
  Other Names: IL-11; Neumega

SUMMARY:
The goal of this clinical research study is to find out if IL-11 (NeumegaTM) may increase the platelet count in patients with Chronic myeloid leukemia (CML) who develop low platelet counts while receiving therapy with imatinib mesylate (Gleevec, STI571), or other tyrosine kinase inhibitors such as AMN107, dasatinib, or SK1606.

Primary Objective:

1. To determine efficacy of low-dose interleukin-11, (IL-11, oprelvekin, NeumegaTM) in improving the thrombocytopenia associate with imatinib or other tyrosine kinase inhibitor therapy in patients with CML.

Secondary Objective:

1. To determine the safety of low-dose IL-11 in patients with CML and thrombocytopenia associated with imatinib or other tyrosine kinase inhibitors

DETAILED DESCRIPTION:
IL-11 is a hormone normally produced in your body that plays a role in stimulating the production of platelets.

Before you can start treatment on this study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will have a blood sample (1 teaspoon) collected to check your platelet count. Women who are able to have children must have a negative blood pregnancy test.

If you are found to be eligible to take part in this study, you will receive one injection of IL-11 under the skin (usually of the arms, legs or abdomen) 3 times a week. If your platelet count increases, treatment will continue on this schedule as long as a platelet increase is observed. If the treatment is well tolerated but there is not enough of a platelet improvement, the dose and frequency of IL-11 injections may be increased. If the platelet count becomes high enough, treatment may be stopped but may also be restarted if necessary.

During therapy with IL-11, additional blood samples (1 teaspoon each) will be collected to measure the platelet count every week until the platelets are stable and then every 2 to 6 weeks while you are receiving treatment on study. No other tests are required for this study.

While you are on this study, you will continue your treatment with imatinib mesylate or other tyrosine kinase inhibitor as decided by your doctor for standard care.You will be taken off if there is no response to treatment or if there are unacceptable side effects. There will be no follow-up after you go off study.

This is an investigational study. The Food and Drug Administration (FDA) has approved IL-11 for use in chemotherapy-caused low platelet counts. A maximum of 30 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* CML patients in chronic or accelerated phase receiving treatment with imatinib mesylate (Gleevec), or other tyrosine kinase inhibitors such as AMN107, dasatinib, or SK1606.
* Grade >/= 3 thrombocytopenia (platelets <50 * 10(9)/L) after the first 4 weeks of therapy with the tyrosine kinase inhibitor. Thrombocytopenia must be either recurrent (i.e., second or greater episode of grade >/= 3 thrombocytopenia) or having required dose reductions of the tyrosine kinase inhibitor.
* Signed informed consent.
* Expected to have therapy with imatinib continued for > 3 months.

Exclusion Criteria:

* Known allergies to E. coli.
* New York Heart Association (NYHA) class III or IV.
* Patient has known hypersensitivity to Neumega or any component of Neumega.
* Thrombocytopenia that is considered to be unrelated to treatment with imatinib.
* Stem cell transplantation within 60 days.
* History of atrial arrhythmias
* Pregnancy
* Papilledema

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E. Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 10/15/05 to 9/17/07. All participants registered at The University of Texas M.D. Anderson Cancer Center.
Period: Overall Study
Arm/Group | Interleukin-11
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Interleukin-11
Number analyzed (Participants) | 8
Age Continuous [Median (Full Range); unit: years] | 55 [31 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response
Description: Number of participants with platelet response of 'Complete Response' (CR) defined as a sustained (>/= 3 months) platelet count >/= 60 x 10^9/L while continuing tyrosine kinase inhibitor (TKI) therapy or sustained (>/= 3 months) re-escalation of TKI dose to the pre-thrombocytopenia level without recurrence of thrombocytopenia.
Time Frame: Weekly platelet count till stabilized with on-going review while receiving treatment (study total 2 years)
Measure: Number; unit: Participants
Arm/Group | Interleukin-11
Number analyzed (Participants) | 8
Participants | 3

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Interleukin-11
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interleukin-11 (N=8)
Edema (General disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Blurry Vision (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes